CLINICAL TRIAL: NCT06139419
Title: A Prospective Phase II Controlled Study to Evaluate the Impact of Thymosin Alpha 1 on the Completion Rate of Consolidation Immunotherapy After Radical Radiochemotherapy for Locally Advanced Non-Small Cell Lung Cancer
Brief Title: The Impact of Thymosin α-1 on the Efficacy of Concurrent Chemoradiotherapy Followed by Immunotherpay Consolidation for Locally Advanced NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-1098
Record Dates: First submitted 2023-08-30; First posted 2023-11-18 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non-small cell lung cancer; Thymosin alpha-1; concurrent chemoradiotherpay; immunotherapy consolidation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Albumin-Bound Paclitaxel; Cisplatin; tislelizumab; Thymalfasin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concurrent Tα-1 group (Experimental): In this concurrent Tα-1 group, participants receive concurrent chemoradiotherapy followed by immunotherapy consolidation. During this treatment, thymosin alpha-1 was administered at 4.8mg each time.
  Interventions: Radiation: definitive radiotherapy; Drug: induction chemo-immunotherapy; Drug: concurrent chemotherapy; Drug: Immunotheapy consolidation; Drug: Thymosin Alpha1
- Control group (Other): In control group, participants receive concurrent chemoradiotherapy followed by immunotherapy consolidation.
  Interventions: Radiation: definitive radiotherapy; Drug: induction chemo-immunotherapy; Drug: concurrent chemotherapy; Drug: Immunotheapy consolidation

INTERVENTIONS:
Radiation: definitive radiotherapy — Participants were treated with definitive thoracic radiotherapy
Drug: induction chemo-immunotherapy — All participants receive two cycles of albumin-bound paclitaxel (260mg/m2) on d1 and cisplatin (25mg/m2) from d1 to d3 in combination with tislelizumab (200mg) on d1.
  Other Names: albumin-bound paclitaxel; cisplatin; tislelizumab
Drug: concurrent chemotherapy — Concurrent chemotherapy consists of weekly albumin-bound paclitaxel (50mg/m2) and cisplatin (25mg/m2).
  Other Names: albumin-bound paclitaxel; cisplatin
Drug: Immunotheapy consolidation — Participants without disease progression, grade ≥3 toxicities, and/or grade ≥2 pneumonitis after CCRT receive tislelizumab 200 mg (Q3W) for up to 12 months.
  Other Names: tislelizumab
Drug: Thymosin Alpha1 — Participants in the Tα1 treatment group will receive Tα1 from the beginning of induction chemo-immunotherapy until the completion of immunotherapy consolidation. In detail, Tα-1 would be administered according to the following three stages:
  1. Induction chemo-immunotherapy: Tα-1 will be subcutaneously administered at 4.8 mg on d1 and d3 for each cycle.
  2. Concurrent chemoradiotherapy: Tα-1 will be subcutaneously administered at 4.8mg biweekly.
  3. Immunotherpay consolidation: Tα-1 will be administered concurrently with tislelizumab at 4.8mg (Q3W) for up to 12 months.
  Other Names: thymalfasin
  Arms: Concurrent Tα-1 group

SUMMARY:
This prospective phase II randomized study is to determine the impact of thymosin alpha-1 on the concurrent chemoradiotherpay followed by immunotherapy consolidation in patients with locally advanced NSCLC by assessing the survival outcomes, treatment responses and toxicities.

DETAILED DESCRIPTION:
This prospective phase II randomized study is to determine the impact of thymosin alpha-1 on the concurrent chemoradiotherpay followed by immunotherapy consolidation in patients with locally advanced NSCLC by assessing the survival outcomes, treatment responses and toxicities.

Patients with locally advanced NSCLC who will receive concurrent radiochemotherapy followed by immunotherapy consolidation will be randomly divided into two groups (concurrent Tα1 treatment group and control group [in which Tα1 will not be used]), and the overall survivals, progression-free survivals (PFS), completion rate of immunotherapy consolidation, toxicities/adverse effects, and peripheral blood immune biomarkers will be compared between these two groups.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years old
* histologically confirmed locally advanced and unresectable NSCLC;
* no prior radiotherapy or surgery;
* with the life expectancy over 12 weeks;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* adequate bone marrow and hepatic and renal functions;
* informed consent

Exclusion Criteria:

* Concurrent enrollment in another clinical trial, unless it is an observational (non-interventional) clinical study;
* With histologically documented combined small-cell lung carcinoma;
* Major surgery (excluding vascular access placement) within 4 weeks prior to enrollment in the study;
* Active or prior documented autoimmune disease within the past 2 years;
* Active or prior documented inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis);
* History of innate immunodeficiency;
* History of organ transplant that requires the use of immunosuppressives;
* A mean heart rate-corrected QT interval (QTc) ≥ 470 ms, calculated using Bazett correction from 3 ECG calculation cycles;
* Poorly managed health conditions that include but are not limited to persistent or active infections, symptomatic congestive heart failure, poorly controlled hypertension, unstable angina, arrhythmia, active peptic ulcer disease or gastritis, active hemorrhagic diseases, hepatitis C or human immunodeficiency virus (HIV) infection, hepatitis B (positive HBsAg and HBV DNA > 500 IU/ml), and mental disorders/social conditions that may hinder the compliance with the study requirements or the ability to give written informed consent willingly;
* Active tuberculosis;
* Receipt of live or attenuated vaccination within 30 days prior to the first dose of the investigational agents;
* History of another primary malignancy within the past 5 years, excluding adequately treated basal or squamous cell skin cancers or cervical carcinoma in situ;
* Pregnant/breastfeeding women or males/females of reproductive potential who do not use contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Completion rate of immunotherapy | Calculated from the start of treatment to one year after the last treatment completion
  Proportion of participants completing 12 months of consolidation of immutherapy

SECONDARY OUTCOMES:
Overall survival | 2 years
Progression-free survival | one year
Incidence of ≥grade 2 pneumonia | through study completion, an average of 1 year
Drop-out rate during the I/O consolidation | One year
The absolute count of total lymphocyte in peripheral blood | Calculated from the start of treatment to one year after the last treatment completion; up to 18 months
  Measured at baseline, before immunotherapy, and every 3-4 months thereafter until the end of immunotherapy.
The expression of peripheral blood cytokines (including IL2, IL4, IL6, IL10, TNF-α, and IFN-γ) | Calculated from the start of treatment to one year after the last treatment completion; up to 18 months
  Measured at baseline, before immunotherapy, and every 3-4 months thereafter until the end of immunotherapy.
The absolute count of peripheral blood lymphocyte subsets (including CD3+, CD3+CD4+, CD3+CD8+, CD19+, CD3-CD16+CD56+, and CD56+ NK cells, PD-1+CD8+ T cells, Tim3+ CD8+ T cells, CD62lowCD4+ T cells, PD-1+CD4+ T cells, and Tim3+CD4+ T cells | Calculated from the start of treatment to one year after the last treatment completion; up to 18 months
  Measured at baseline, before immunotherapy, and every 3-4 months thereafter until the end of immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Professor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun yat-sen university cancer center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spigel DR, Faivre-Finn C, Gray JE, Vicente D, Planchard D, Paz-Ares L, Vansteenkiste JF, Garassino MC, Hui R, Quantin X, Rimner A, Wu YL, Ozguroglu M, Lee KH, Kato T, de Wit M, Kurata T, Reck M, Cho BC, Senan S, Naidoo J, Mann H, Newton M, Thiyagarajah P, Antonia SJ. Five-Year Survival Outcomes From the PACIFIC Trial: Durvalumab After Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. J Clin Oncol. 2022 Apr 20;40(12):1301-1311. doi: 10.1200/JCO.21.01308. Epub 2022 Feb 2. PMID 35108059
- [Background] Yegya-Raman N, Friedes C, Sun L, Iocolano M, Kim KN, Doucette A, Cohen RB, Robinson KW, Levin WP, Cengel KA, Lally B, Agarwal M, D'Avella CA, Marmarelis ME, Kosteva JA, Singh AP, Ciunci CA, Aggarwal C, Berman AT, Langer CJ, Feigenberg SJ. Utilization and Factors Precluding Receipt of Checkpoint Inhibitor Consolidation for Stage III NSCLC in a Large US Academic Health System. Clin Lung Cancer. 2023 Jul;24(5):474-482. doi: 10.1016/j.cllc.2023.03.013. Epub 2023 Apr 3. PMID 37076396
- [Background] Bryant AK, Yin H, Schipper MJ, Paximadis PA, Boike TP, Bergsma DP, Movsas B, Dess RT, Mietzel MA, Kendrick R, Seferi M, Dominello MM, Matuszak MM, Jagsi R, Hayman JA, Pierce LJ, Jolly S; Michigan Radiation Oncology Quality Consortium. Uptake of Adjuvant Durvalumab After Definitive Concurrent Chemoradiotherapy for Stage III Nonsmall-cell Lung Cancer. Am J Clin Oncol. 2022 Apr 1;45(4):142-145. doi: 10.1097/COC.0000000000000899. PMID 35271524
- [Background] Wu J, Zhou L, Liu J, Ma G, Kou Q, He Z, Chen J, Ou-Yang B, Chen M, Li Y, Wu X, Gu B, Chen L, Zou Z, Qiang X, Chen Y, Lin A, Zhang G, Guan X. The efficacy of thymosin alpha 1 for severe sepsis (ETASS): a multicenter, single-blind, randomized and controlled trial. Crit Care. 2013 Jan 17;17(1):R8. doi: 10.1186/cc11932. PMID 23327199
- [Background] Romani L, Bistoni F, Gaziano R, Bozza S, Montagnoli C, Perruccio K, Pitzurra L, Bellocchio S, Velardi A, Rasi G, Di Francesco P, Garaci E. Thymosin alpha 1 activates dendritic cells for antifungal Th1 resistance through toll-like receptor signaling. Blood. 2004 Jun 1;103(11):4232-9. doi: 10.1182/blood-2003-11-4036. Epub 2004 Feb 24. PMID 14982877
- [Background] Liu F, Qiu B, Xi Y, Luo Y, Luo Q, Wu Y, Chen N, Zhou R, Guo J, Wu Q, Xiong M, Liu H. Efficacy of Thymosin alpha1 in Management of Radiation Pneumonitis in Patients With Locally Advanced Non-Small Cell Lung Cancer Treated With Concurrent Chemoradiotherapy: A Phase 2 Clinical Trial (GASTO-1043). Int J Radiat Oncol Biol Phys. 2022 Nov 1;114(3):433-443. doi: 10.1016/j.ijrobp.2022.07.009. Epub 2022 Jul 21. PMID 35870709
- [Background] Garaci E, Pica F, Serafino A, Balestrieri E, Matteucci C, Moroni G, Sorrentino R, Zonfrillo M, Pierimarchi P, Sinibaldi-Vallebona P. Thymosin alpha1 and cancer: action on immune effector and tumor target cells. Ann N Y Acad Sci. 2012 Oct;1269:26-33. doi: 10.1111/j.1749-6632.2012.06697.x. PMID 23045967
- [Background] Wara WM, Ammann AJ, Wara DW. Effect of thymosin and irradiation on immune modulation in head and neck and esophageal cancer patients. Cancer Treat Rep. 1978 Nov;62(11):1775-8. PMID 728896
- [Background] Danielli R, Cisternino F, Giannarelli D, Calabro L, Camerini R, Savelli V, Bova G, Dragonetti R, Di Giacomo AM, Altomonte M, Maio M. Long-term follow up of metastatic melanoma patients treated with Thymosin alpha-1: investigating immune checkpoints synergy. Expert Opin Biol Ther. 2018 Jul;18(sup1):77-83. doi: 10.1080/14712598.2018.1494717. PMID 30063847